CLINICAL TRIAL: NCT01245738
Title: Dyslipidemia: REsidual and Mixed Abnormalities IN Spite of Statin Therapy: The Dyslipidemia REMAINS Study: A Multicenter, Prospective, Observational Study of Lipid Profiles and Treatment Patterns at Presentation and After 12 Weeks of Statin Therapy Among Indian Adults Presenting With First Coronary Event
Brief Title: Effect of Statins on Lipid Levels Following the First Acute Coronary Event (MK-0000-204)
Acronym: REMAINS
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0000-204; CTRI/2013/02/003429 (Registry Identifier: CTRI)
Record Dates: First submitted 2010-08-13; First posted 2010-11-22 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Dyslipidemias; Hypercholesterolemia; Hypertriglyceridemia; High LDL-C; Low HDL-C
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia; Hypertriglyceridemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants: Participants admitted to participating tertiary cardiac care centers who experienced a first coronary event.

SUMMARY:
The current study is proposed to investigate the pattern of dyslipidemia and of lipid treatment practices in patients in India experiencing their first acute cardiovascular event and the extent of residual dyslipidemia after 12 weeks of treatment with statins. Dyslipidemia definitions are per the National Cholesterol Education Program - Adult Treatment Panel III (NCEP-ATP III).

ELIGIBILITY:
Inclusion Criteria:

* Currently admitted with a confirmed diagnosis of first acute coronary event (STEMI/NSTEMI/Unstable Angina)
* Access to medical records covering the entire study period, and availability of data required for the study
* Potential to collect blood sample within 24 hours of onset for symptoms
* Considered for initiation/maintenance/modification of statin therapy before discharge from hospital
* Willing to comply with the study requirements

Exclusion Criteria:

* Participating in a clinical trial or any type of other clinical study involving therapeutic intervention or otherwise failing to consent to interview
* Known inherited disorder of lipoprotein metabolism
* History of hypothyroidism, nephrotic syndrome, chronic alcoholism, Cushing syndrome

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients experiencing their first acute coronary event who are admitted to participating tertiary cardiac care centers in India will potentially be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 635 (Actual)
Dates: Start 2010-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0000-204&kw=0000-204&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data were collected at the time of the first acute coronary event and 12 weeks after post-event statin therapy among participants across 19 tertiary cardiac care centers in India.
Pre-assignment Details: 635 participants were considered eligible for the study, however; only 514 started (had complete baseline data).
Period: Overall Study
Arm/Group | Participants
Started | 514
Completed | 474
Not Completed | 40

BASELINE CHARACTERISTICS:
Population: Participants admitted to participating tertiary cardiac care centers who experienced a first coronary event.
Arm/Group | Participants
Number analyzed (Participants) | 474
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94
  Male | 380

OUTCOME MEASURES:

1. Primary Outcome: Total Cholesterol (TC) Levels at First Acute Coronary Event
Description: At the time of hospital admission for a first acute coronary event, the TC levels of eligible participants were taken. This level was considered the baseline value. A TC level of >240 mg/dL is considered an abnormal lipid value (dyslipidemia).
Time Frame: At hospital presentation (Day 1)
Population: Participants who had a total cholesterol measurement at baseline.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Participants
Number analyzed (Participants) | 474
mg/dL | 163.5 (42.16)

2. Primary Outcome: Low-Density Lipoprotein Cholesterol (LDL-C) Levels at First Acute Coronary Event
Description: At the time of hospital admission for a first acute coronary event, the LDL-C levels of eligible participants were taken. This level was considered the baseline value. A LDL-C level of >70 mg/dL is considered an abnormal lipid value (dyslipidemia).
Time Frame: At hospital presentation (Day 1)
Population: Participants who had a LDL-C measurement at baseline.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Participants
Number analyzed (Participants) | 472
mg/dL | 105.9 (37.55)

3. Primary Outcome: High-Density Lipoprotein Cholesterol (HDL-C) Levels at First Acute Coronary Event
Description: At the time of hospital admission for a first acute coronary event, the HDL-C levels of eligible participants were taken. This level was considered the baseline value. A HDL-C level of <40 mg/dL is considered an abnormal lipid value (dyslipidemia).
Time Frame: At hospital presentation (Day 1)
Population: Participants who had a HDL-C measurement at baseline.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Participants
Number analyzed (Participants) | 474
mg/dL | 42.9 (17.23)

4. Primary Outcome: Triglycerides (TG) Levels at First Acute Coronary Event
Description: At the time of hospital admission for a first acute coronary event, the TG levels of eligible participants were taken. This level was considered the baseline value. A TG level of >150 mg/dL is considered an abnormal lipid value (dyslipidemia).
Time Frame: At hospital presentation (Day 1)
Population: Participants who had a TG measurement at baseline.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Participants
Number analyzed (Participants) | 474
mg/dL | 146.9 (97.65)

5. Primary Outcome: Change From Baseline in TC Levels After Treatment
Description: TC levels were measured after 12 weeks of treatment with a statin. The change from baseline was calculated as the difference between baseline and Week 12 values.
Time Frame: Baseline and at Week 12
Population: Participants of the Full Analysis Set (FAS) Population who had a TC measurements at baseline and Week 12.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Participants
Number analyzed (Participants) | 471
mg/dL | -32.2 (48.56)

6. Primary Outcome: Change From Baseline in LDL-C Levels After 12 Weeks of Treatment With Statins
Description: LDL-C levels were measured after 12 weeks of treatment with a statin. The change from baseline was calculated as the difference between baseline and Week 12 values.
Time Frame: Baseline and at Week 12
Population: Participants of the FAS Population who had LDL-C measurements at baseline and Week 12.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Participants
Number analyzed (Participants) | 468
mg/dL | -32.2 (42.57)

7. Primary Outcome: Change From Baseline in HDL-C Levels After 12 Weeks of Treatment With Statins
Description: HDL-C levels were measured after 12 weeks of treatment with a statin. The change from baseline was calculated as the difference between baseline and Week 12 values.
Time Frame: Baseline and at Week 12
Population: Participants of the FAS Population who had HDL-C measurements at baseline and Week 12.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Participants
Number analyzed (Participants) | 471
mg/dL | -1.2 (18.01)

8. Primary Outcome: Change From Baseline in TG Levels After 12 Weeks of Treatment With Statins
Description: TG levels were measured after 12 weeks of treatment with a statin. The change from baseline was calculated as the difference between Baseline and Week 12 values.
Time Frame: Baseline and at Week 12
Population: Participants of the FAS Population who had TG measurements at baseline and Week 12.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Participants
Number analyzed (Participants) | 471
mg/dL | 1.6 (97.26)

9. Primary Outcome: Percentage of Participants Who Achieved Target Lipid Levels for LDL-C But Did Not Achieve Target Lipid Levels for HDL-C and TG After 12 Weeks of Treatment With Statins
Description: The percentage of participants who achieved predefined lipid target levels after 12 weeks of treatment with statins. Predefined lipid target levels were: LDL-C less than 70 mg/dL, HDL-C greater than 40 mg/dL, and TG less than 150 mg/dL.
Time Frame: Week 12
Population: Participants of the FAS Population who had HDL-C, TG, and LDL-C measurements at Week 12.
Measure: Number; unit: Percentage of Participants
Arm/Group | Participants
Number analyzed (Participants) | 474
Percentage of Participants | 11.6

10. Primary Outcome: Percentage of Participants Who Achieved Target Lipid Levels for TG and LDL-C But Did Not Achieve Target Lipid Levels for HDL-C After 12 Weeks of Treatment With Statins
Description: as for outcome 9
Time Frame: Week 12
Population: Participants of the FAS Population who had HDL-C, TG, and LDL-C measurements and Week 12.
Measure: Number; unit: Percentage of Participants
Arm/Group | Participants
Number analyzed (Participants) | 474
Percentage of Participants | 54.4

11. Primary Outcome: Percentage of Participants Who Achieved Target Lipid Levels of HDL-C and LDL-C But Did Not Achieve Target Lipid Levels for TG After 12 Weeks of Treatment With Statins
Description: as for outcome 9
Time Frame: Week 12
Population: Participants of the FAS Population who had HDL-C, TG, and LDL-C measurements and Week 12.
Measure: Number; unit: Percentage of Participants
Arm/Group | Participants
Number analyzed (Participants) | 474
Percentage of Participants | 17.1

12. Primary Outcome: Percentage of Participants Who Did Not Achieve Target Lipid Levels for LDL-C, HDL-C, and TG After 12 Weeks of Treatment With Statins
Description: as for outcome 9
Time Frame: Week 12
Population: Participants of the FAS Population who had HDL-C, TG, and LDL-C measurements and Week 12.
Measure: Number; unit: Percentage of Participants
Arm/Group | Participants
Number analyzed (Participants) | 474
Percentage of Participants | 1.1

13. Primary Outcome: Percentage of Participants Who Achieved Target Lipid Levels for TG But Did Not Achieve Target Lipid Levels for HDL-C and LDL-C After 12 Weeks of Treatment With Statins
Description: as for outcome 9
Time Frame: Week 12
Population: Participants of the FAS Population who had HDL-C, TG, and LDL-C measurements and Week 12.
Measure: Number; unit: Percentage of Participants
Arm/Group | Participants
Number analyzed (Participants) | 474
Percentage of Participants | 1.3

14. Primary Outcome: Percentage of Participants Who Achieved Target Lipid Levels of HDL-C But Did Not Achieve Target Lipid Levels for TG and LDL-C After 12 Weeks of Treatment With Statins
Description: as for outcome 9
Time Frame: Week 12
Population: Participants of the FAS Population who had HDL-C, TG, and LDL-C measurements and Week 12.
Measure: Number; unit: Percentage of Participants
Arm/Group | Participants
Number analyzed (Participants) | 474
Percentage of Participants | 0.6

ADVERSE EVENTS:
Time Frame: Up to 12 Weeks
Arm/Group | Participants
Serious Adverse Events (participants affected / at risk) | 6/474
Other Adverse Events (participants affected / at risk) | 0/474
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants (N=474)
Coronary artery disease (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 4 (4)
Gastroenteritis (Infections and infestations) | 1 (1)
Sensory Disturbance (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The scientific information generated from this study will be publically disclosed in forms of peer reviewed publication and scientific presentations and may even be actively disseminated amongst the practicing medical community in appropriate scientific platforms.